CLINICAL TRIAL: NCT00796523
Title: A Randomized, Controlled Trial to Decrease Infant Crying
Brief Title: An Intervention to Decrease Infant Crying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riverside Methodist Hospital (Other)
Collaborators: Prevent Child Abuse America (Unknown)
Responsible Party: Jonna M. McRury, M.D., University of Toledo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 941
Record Dates: First submitted 2008-10-16; First posted 2008-11-24 (Estimated); Results first posted 2008-11-24 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Colic
Keywords: colic; crying; clinical trial
MeSH Terms: conditions — Colic; Crying

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Happiest Baby videotape (Experimental): videotape describing the Happiest Baby on the Block technique
  Interventions: Behavioral: Happiest Baby videotape
- control videotape (Placebo Comparator): videotape with normal newborn instruction
  Interventions: Behavioral: control videotape

INTERVENTIONS:
Behavioral: Happiest Baby videotape — a videotape demonstrating the Happiest Baby on the Block technique for calming crying infants
  Other Names: Happiest Baby on the Block technique
  Arms: Happiest Baby videotape
Behavioral: control videotape — a videotape with general newborn care instructions
  Other Names: Civitas' Begin with Love
  Arms: control videotape

SUMMARY:
This is a study looking at the Happiest Baby on the Block technique. The investigators hypothesized that infants of mothers given a 30 minute videotape demonstrating the Happiest Baby on the Block technique would fuss/cry less and sleep longer than infants of mothers given a 30 minute videotape on general newborn care. The investigators also hypothesized that mothers given the Happiest Baby on the Block videotape would have lower levels of stress.

DETAILED DESCRIPTION:
Mothers recorded their babies fussing, crying and sleeping on paper diaries when their infants were 1, 4, 6, 8 and 12 weeks old.

ELIGIBILITY:
Inclusion Criteria:

Mothers of singleton newborns

* 37 to 41 week gestation
* healthy (no ICU admission)

Exclusion Criteria:

* not able to view videotape at home
* not able to speak English

Max Age: 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2005-08; Primary Completion 2006-02 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonna M. McRury, M.D., Principal Investigator — University of Toledo
Locations (1):
- Riverside Methodist Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers of healthy singleton newborn infants with a gestational age of 37-41 weeks admitted to the normal newborn nursery of a large community hospital were given a flier inviting them to participate by contacting the research assistant by phone.
Pre-assignment Details: 1408 Fliers were distributed and 51 mothers contacted the research assistant for enrollment in the study.
Period: Overall Study
Arm/Group | Happiest Baby Videotape | Control Videotape
Started | 27 | 24
Completed | 18 | 17
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Happiest Baby Videotape | Control Videotape | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Categorical [Count of Participants; unit: Participants] — (mothers)
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 27 | 24 | 51
    >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — (mothers)
  years | 29 (6) | 30 (4) | 29 (5)
Age Continuous [Mean (Standard Deviation); unit: days] — (babies)
  days | 3 (1) | 3 (1) | 3 (1)
Age, Customized [Number; unit: participants] — (babies)
  participants
    <=5 days | 27 | 24 | 51
    >5 days | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 51

OUTCOME MEASURES:

1. Secondary Outcome: Parenting Stress Index
Description: a continuous scale measuring stress with a range of 131 (low) to 320 (high); the average person's stress scores are between 188 and 252.
Time Frame: week 6
Population: results based on ITT; 16 subjects did not complete any diaries or data collection instruments and are not included in the analysis
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Happiest Baby Videotape | Control Videotape
Number analyzed (Participants) | 18 | 17
points on a scale | 225.3 (35.3) | 188.9 (27.9)

2. Primary Outcome: Hours Per Day of Fuss/Cry
Description: total hours per day of fuss, cry, and unsoothable crying.
Time Frame: week 8
Population: If fewer than 3 diaries were completed for a given time period (that is, one or two of the days was missing or had more than 180 minutes unrecorded), then the average of only the completed diaries was used. Results are based on ITT; 16 subjects did not complete any diaries and are not included in the analysis
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Happiest Baby Videotape | Control Videotape
Number analyzed (Participants) | 18 | 17
hours per day | 2.20 (1.25) | 1.48 (1.23)

3. Primary Outcome: Hours Per Day of Sleep
Description: mean sleep time is the mean of 3 daily sleep times reported in a time period.
Time Frame: week 8
Population: Results based on ITT; 16 subjects did not complete any diaries and are not included in the analysis
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Happiest Baby Videotape | Control Videotape
Number analyzed (Participants) | 18 | 17
hours per day | 13.87 (1.60) | 14.1 (1.73)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No